CLINICAL TRIAL: NCT05692908
Title: An Open-Label, Dose-Escalation Study of the Safety of an Anti-CD38 Antibody Drug Conjugate (STI-6129) in Patients With Relapsed or Refractory Systemic AL Amyloidosis
Brief Title: An Open-Label Study of the Safety of an Anti-CD38 Antibody Drug Conjugate (STI-6129) in Patients With AL Amyloidosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sorrento Therapeutics filed for chapter 11 bankruptcy.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 38ADC-RRAL-102-SWE
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Light Chain (AL) Amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STI-6129 infusion (Experimental): Intravenous infusion to be given with prophylaxis for infusion reactions if necessary.
  Interventions: Biological: STI-6129

INTERVENTIONS:
Biological: STI-6129 — Four cycles of intravenous infusion of STI-6129 will be given (one infusion every four weeks).
  Other Names: anti-CD38-Duostatin 5.2 antibody-drug conjugate (ADC)

SUMMARY:
This is a Phase 1 open-label, dose escalation trial designed to identify the recommended phase 2 dose of STI-6129 by assessing the safety, preliminary efficacy, and immunogenicity in subjects with relapsed or refractory systemic AL Amyloidosis

DETAILED DESCRIPTION:
This study is an open-label, dose-finding, to identify the recommended phase 2 dose (RP2D) of STI-6129 by assessing the safety, and pharmacokinetics for the treatment of RRAL which is defined as the development of disease progression during therapy with an anti-AL amyloidosis treatment regimen or within 60 days of the last dose of an anti-AL amyloidosis treatment regimen or the achievement of less than a PR after ≥ 2 cycles.

The trial is the dose-escalation study. A standard dose escalation 3+3 will be utilized to identify dose-limiting toxiticy (DLTs) and a safe maximum tolerated dose (MTD) of STI-6129 in patients with R/R systemic AL amyloidosis. A total of 6 dosing cohorts are planned from 0.88 mg/kg to 3.68 mg/kg. Approximate dosing increments between cohorts are 1.33x up to the maximum planned dose level.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years.
* 2. Confirmed diagnosis of AL amyloidosis by tissue biopsy of an involved organ, or a surrogate site such as abdominal fat, demonstrating amyloid deposition by mass spectrometry
* 3. The presence of a monoclonal light chain protein in serum and/or urine
* 4. Relapsed or refractory (R/R) AL amyloidosis is patients who have exhausted standard of care treatment. Patients who have received prior CD38-directed monoclonal antibody (e.g. daratumumab, isatuximab) treatment or prior stem cell transplantation remain eligible. Patients may have relapsed with disease progression or have been refractory to their last prior line of treatment. Refractory systemic AL amyloidosis is defined as the development of disease progression during therapy with an anti-AL amyloidosis treatment regimen or within 60 days of the last dose of an anti-AL amyloidosis treatment regimen or the achievement of less than a PR after ≥ 2 cycles
* 5. Measurable disease defined by the following: the finding by serum FLC assay that the difference between the involved and uninvolved FLC (dFLC) is ≥ 40 mg/L
* 6. Pulse oximetry ≥ 92% on room air
* 7. ECOG performance status of 0, 1, or 2
* 8. Be willing and able to comply with the study schedule and all other protocol requirements
* 9. Willing to follow contraception guidelines: c. If a female, be sterile (surgically or biologically)* or at least one year post-menopausal, or have a monogamous partner who is surgically sterile, or have a same sex partner, or if in a heterosexual relationship, must agree to do the following during the study after completing IP dosing:

  * Practice abstinence (only considered an acceptable method of contraception when it is in line with the participants' usual and preferred lifestyle)
  * Use at least one of the following medically acceptable methods of birth control:
* Hormonal methods as follows:

  * Combined estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  * Progestogen only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* Intrauterine devices
* Intrauterine hormone-releasing systems
* Vasectomized partner
* Barrier contraception

  * Defined as having had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; or having a congenital or acquired condition that prevents childbearing.

    d. If a male of reproductive potential, unless he has a same sex partner, must agree to do the following during the study after completing IP dosing:
    * Refrain from donating sperm
    * Practice abstinence from heterosexual activity (only considered an acceptable method of contraception when it is in line with the participants' usual and preferred lifestyle), OR
    * Use (or have their partner use) acceptable contraception (see criterion above) during heterosexual activity, such as barrier contraception

Exclusion Criteria:

* 1. Isolated vascular amyloid in a bone marrow biopsy or a plasmacytoma specimen or isolated soft tissue involvement (localized AL amyloidosis)
* 2. Presence of non-AL amyloidosis
* 3. A diagnosis of multiple myeloma
* 4. A diagnosis of other malignancies if the malignancy has required therapy within the last 3 years or is not in complete remission. Exceptions are non-metastatic basal cell or squamous cell carcinomas of the skin or prostate cancer or in situ cancer that does not require treatment or is well under control
* 5. Treatment with an allogeneic hematopoietic stem cell transplantation (HSCT) within 6 months prior to the planned infusion of STI-6129, or active graft-versus-host disease (GvHD) following the allogeneic transplant, or a requirement for currently receiving immunosuppressive therapy following the allogeneic transplant
* 6. Revised Mayo Clinic AL amyloidosis stage > 3
* 7. New York Heart Association (NYHA) class > 3
* 8. Left ventricular ejection fraction (LVEF) < 40%.
* 9. Patients with mean left ventricular wall thickness ≥ 15 mm and/or intraventricular septal thickness > 25 mm by echocardiogram in the absence of hypertension or valvular heart disease
* 10. Patients with NT-proBNP ≥ 1800 ng/L or BNP ≥ 400 ng/L, cTnT ≥ 0.025 mcg/L will be excluded in the dose-escalation stage of the study and can only be included in the PK and expansion stages after evaluation by cardiology and discussion with the principle investigator regarding the risk associated with the treatment
* 11. The following baseline hematological laboratory results at Screening (these results must be independent of blood product or hematopoietic growth factor support):

  1. Hemoglobin < 8.0 g/dL
  2. Platelet count < 50,000/μL
  3. Absolute neutrophil count (ANC) < 1000/ μL
* 12. The following baseline chemistry laboratory results at Screening:

  1. Serum creatinine > 2.0 x the upper limit of normal (ULN), or estimated creatinine clearance < 45 mL/min (using the Cockcroft-Gault equation).
  2. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x ULN or serum total bilirubin > 1.5x ULN (except for patients in whom hyperbilirubinemia is attributed to Gilbert's Syndrome)
* 13. INR or aPTT > 1.5x ULN within 1 week prior to the infusion of STI-6129, unless on a stable dose of an anticoagulant
* 14. Are pregnant or breastfeeding
* 15. Patients with ≥ Grade 3 neuropathy or Grade 2 neuropathy with associated pain
* 16. Active bacterial, viral, or fungal infection within 72 hours of the infusion of STI-6129; patients with ongoing use of prophylactic antibiotics, antifungal agents, or antiviral agents remain eligible as long as there is no evidence of active infection, or the STI-6129 treatment would put the patient at risk for a meaningful safety event.
* 17. Have a prolongation in QTcF (Fridericia correction formula) > 480 msec on a baseline ECG
* 18. Any condition including the presence of laboratory abnormalities that places the patient at an unacceptable risk if the patient was to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Safety of STI-6129 | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of adverse events (AEs), severe AEs (SAEs), DLTs, neurotoxicity and laboratory abnormalities using the Common Terminology Criteria for Adverse Events (CTCAE Version 5)

SECONDARY OUTCOMES:
Overall hematological response rate according to the 2012 Consensus Round Table response criteria | Baseline through study completion at up to approximately 24 months
  Proportion of subjects with Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), No Response (NR) and Progressive Disease (PD)
Organ response rates (cardiac, renal, hepatic, peripheral nervous system) according to the 2012 Consensus Round Table response criteria | Baseline through study completion at up to approximately 24 months
  Organ response rates (cardiac, renal, hepatic, peripheral nervous system) according to the 2012 Consensus Round Table response criteria
Correlation of treatment response (organ responses and hematological response) with disease severity based on the 2012 revised Mayo Clinic staging system for AL amyloidosis | Baseline through study completion at up to approximately 24 months
  Correlation of treatment response (organ responses and hematological response) with disease severity based on the 2012 revised Mayo Clinic staging system for AL amyloidosis
Plasma levels of the total antibody plus conjugated toxin (STI-6129) and the free toxin (Duostatin 5.2) | Baseline through study completion at up to approximately 24 months
  Plasma levels of the total antibody plus conjugated toxin (STI-6129) and the free toxin (Duostatin 5.2) by ELISA and mass spectrophotometry assays, respectively, at pre-dose and various time points post-dose